CLINICAL TRIAL: NCT04723589
Title: Restoration of Endothelial Integrity in Patients With COVID-19 (RELIC)
Acronym: RELIC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Widespread vaccine availability
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rondi Gelbard, Associate Professor, Department of Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300005853
Record Dates: First submitted 2020-11-26; First posted 2021-01-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Group 1: Standard care for COVID-19 Group 2: Standard care plus non-convalescent plasma infusion
Masking Description: Masking will not be used. Participants randomized to standard care will not receive a sham treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Arm (No Intervention): Participants randomized to standard care will not receive an intervention but will participate in other study procedures, which are blood collection and data collection.
- Intervention Arm (Experimental): Participants randomized to the intervention arm will receive standard care plus an infusion of thawed plasma, starting rate 30 ml/hour for 24 hours, increased to 50 ml/hour if deemed to be hypovolemic (low fluid volume). Only non-convalescent (COVID-antibody-free) plasma will be used.
  Interventions: Biological: Thawed plasma

INTERVENTIONS:
Biological: Thawed plasma — Plasma not labeled "convalescent plasma" is presumed to be free of COVID antibodies, but is not tested for antibodies. To ensure that we are using antibody-free plasma, we will test each unit of plasma with a quick COVID test before it is utilized in this study.
  Arms: Intervention Arm

SUMMARY:
This is a pilot study designed to demonstrate the feasibility of conducting a larger study of standard plasma therapy in COVID-19 patients.

DETAILED DESCRIPTION:
This is a randomized trial in hospitalized COVID-19-positive patients. This trial compares standard care to standard care plus an infusion of non-convalescent thawed plasma. Blood will be collected from all participants at eight timepoints, and clinical data will be collected for 30 days or until discharge/death.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* COVID-19 positive by PCR or assay within 72 hours or less
* Oxygen saturation of ≤94% on room air or requiring supplemental oxygen at screening

Exclusion Criteria:

* mechanically ventilated
* pregnant
* prisoners
* receiving resuscitation with blood products for hemorrhagic shock
* receiving an investigational therapy for COVID-19
* diagnosed with severe comorbidities
* not expected to survive more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants completing plasma infusion for COVID-19 | Track patient progress for 30 days post transfusion.
  Identification of patient population who are COVID-19-positive and transfused with plasma
Number of participants intubated | Track patient progress for 30 days post transfusion
  Participants who are intubated during hospital stay

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score change | Track patient progress for 30 days post transfusion
  SOFA is used as a clinical indicator of morbidity severity. The scale is 0-24, with 0 being normal.
National Early Warning Score change | Track patient progress for 30 days post transfusion
  This score is used as a clinical indicator of patient deterioration. The total possible score ranges from 0 to 20. The higher the score the greater the clinical risk.
Ventilator-free Days | Track patient progress for 30 days post transfusion
  Number of in-hospital days that patient is not ventilated
Intensive care unit-free Days | Track patient progress for 30 days post transfusion
  Number of days patient is hospitalized and not in ICU
In hospital mortality | Track patient progress for 30 days post transfusion
  Number of patients who receive transfusion but do not survive for 30 days
Angiopoietin 1&2 blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  Angiopoietin, a protein, that plays a role in blood vessel formation
Soluble Tie2 blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  Soluble Tie2 is a protein that mediates the function of angiopoietin
Soluble Thrombomodulin blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test indicates blood vessel injury
Syndecan-1 blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test indicates blood vessel injury
Prothrombin time blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test measures blood coagulation
Partial thromboplastin time blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test measures blood coagulation
D-dimer blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test measures for D-dimer concentration, indicating that the blood has been breaking down blood clots
Fibrinogen blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  Tests for a protein important to clotting
Thromboelastography blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  Measures blood coagulation
Von Willebrand Factor Antigen blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test measures a blood clotting protein
Factor VIII blood test | 0, 12, 24, 48, 72 hours. Day 7, 14 and 30.
  This test measures a blood clotting protein

CONTACTS AND LOCATIONS:
Overall Officials: Rondi Gelbard, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No